CLINICAL TRIAL: NCT03913572
Title: Treatment of Perianal Disease Using Adipose-derived Stem Cells
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Samuel.Eisenstein, Prinicipal Investigator, University of California, San Diego
Other Study IDs: 180652
Record Dates: First submitted 2019-02-27; First posted 2019-04-12 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Perianal Fistula; Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- REVOLVE: Patients that have agreed to be prospectively enrolled in the study and undergo Injection of adipose-derived stem cells into perianal fistula with the REVOLVE system
  Interventions: Procedure: Injection of adipose-derived stem cells into perianal fistula
- Retrospective cohort: Patients that have undergone treatment of perianal disease without use of adipose-derived stem cell injection.

INTERVENTIONS:
Procedure: Injection of adipose-derived stem cells into perianal fistula — The plastic surgery team will perform fat graft harvest. Tumescent solution will be infiltrated into the area of liposuction, generally the abdomen, flanks, or thighs. Approximately a00ml of liposuction aspirate will be retrieved. It will be washed and condensed down to about 5-25 ml of good-quality fat graft using the REVOLVE System by Acelity. This will then be loaded into a syringe fitted with an injection cannula. The colorectal surgeon will perform an exam under anesthesia and determine if any additional procedure such as ligation of fistula tract, fistulotomy, endorectal advancement flap, or seton placement/exchange is needed. Severity of disease at time of surgery will be recorded by the attending surgeon. Following any indicated procedure, the lipoaspirate will be injected into the soft tissues around the fistula tract.
  Groups: REVOLVE

SUMMARY:
This study will compare healing and surgical outcomes in patients with chronic perianal disease treated with Adipose-derived Stem Cells (ASCs) to outcomes in patients treated in traditional surgical techniques without ASCs. The study will perform retrospective medical record analysis to clinically characterize patients that have undergone these surgical procedures and compare follow-up data and disease status to determine efficacy of treatment with ASCs compared to similar treatments without the use of ASCs. This will help determine overall efficacy of the treatment as well as determine patient characteristics that may predict treatment success. The study will also prospectively recruit patients with perianal disease that are planning to receive treatment with ASCs, and analyze their outcomes in the same way. Medical record review of outcomes in patients with perianal disease that received treatment with ASCs compared to those that did not will determine efficacy of this procedure.

DETAILED DESCRIPTION:
Specific Aims:

1. Conduct a retrospective review of health information data from patients who have undergone surgery with a colorectal surgery attending at the University of California San Diego, including surgical treatment of perianal fistulas or other chronic perianal diseases, with or without injection of lipoaspirate containing adipose-derived stem cells. Patient data from December 2013 to April 1, 2018, will be obtained, with parameters including date of birth, sex, date of surgery, medical history, surgical history, laboratory values, perioperative data such as blood loss, length of surgery, operative complications, readmissions, and long-term complications and status of disease.
2. Conduct an observational study comparing outcomes of patients that plan to undergo treatment of perianal disease using ASCs compared to those that do not use ASCs. Patients identified as candidates for the procedure by the colorectal surgeons and are planning to undergo the procedure will give informed consent and be recruited into the study. Participants will undergo isolation of ASCs using the REVOLVE ™ System and injection of ASCs into perianal wounds. Clinical data will be analyzed to determine efficacy of the procedure as a means of treating perianal disease.
3. Use the above data to clinically characterize patients that undergo this surgical procedure and what patient characteristics may determine outcomes. Comparing follow-up data and disease status will determine efficacy of treatment with adipose-derived stem cells compared to similar treatments without the use of stem cells.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women, age 18 years of age
2. Diagnosis of perianal disease with tissue defect or chronic wound
3. Underwent, or candidate for, surgery for perianal disease with colorectal surgery attending at UCSD
4. Any ethnic background
5. Any health status
6. Minimum of 30 days postoperative follow-up

Exclusion Criteria:

1. Pregnant women
2. Children less than 18 years old
3. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient's will be identified by colorectal surgeons as those with perianal disease that may benefit from the procedure above. The patients must be able to give consent for the study and complete the Perianal Crohn's Disease Activity Index in English, qualify medically for the surgical procedure, and agree to undergo treatment of perianal disease with injection of lipoaspirate.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2018-09-27 (Actual); Primary Completion 2021-06-26 (Estimated); Study Completion 2021-07-26 (Estimated)

PRIMARY OUTCOMES:
Improvement in perianal disease after the procedure | 4 months
  Patients will have routine post-operative follow up in with a colorectal surgeon and/or their clinical Nurse Practitioner 2-4 weeks following the procedure in colorectal surgery clinic. At that appointment, the timing of additional postoperative appointments or procedures will be determined. Clinical data and status of the disease will be documented by the attending surgeon and subsequently collected from the medical record. Fistula healing will be assessed clinically 3 months after the procedure has been performed. The patient will be asked to complete the Perianal Disease Activity Index (PDAI)questionnaire both prior to intervention as well as at a post-operative appointment 3 months following the procedure to asses for improvement of symptoms. The PDAI is a validated instrument to assess the severity of perianal disease . We will also perform MRIs prior to repair and after to confirm resolution of abscess cavities and fistulae.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Eisenstein, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No